CLINICAL TRIAL: NCT03517137
Title: Very Early PET-response Adapted Targeted Therapy for Advanced Hodgkin Lymphoma: a Single -Arm Phase II Study
Acronym: COBRA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1537-LYMG
Record Dates: First submitted 2018-04-05; First posted 2018-05-07 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Advanced Hodgkin Lymphoma
Keywords: advanced Hodgkin lymphoma; brentuximab vedotin; phase 2
MeSH Terms: interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine; Etoposide; Cyclophosphamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Brentuximab Vedotin; Drug: Adriamycin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Etoposide; Drug: Cyclophosphamide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Brentuximab Vedotin — For PET positive (score of 4-5 following Deauville Criteria) patients: Brentuximab vedotin is administered as an IV infusion over a period of 30 minutes at 1.8 mg/kg on day 1, every 3 weeks (6 cycles); For PET negative (score of 1-3 following Deauville Criteria) patients: Brentuximab vedotin is administered as an IV infusion over a period of 30 minutes at 1.2 mg/kg on day 1 and 15, every 4 weeks (5 cycles)
Drug: Adriamycin — For PET positive (score of 4-5 following Deauville Criteria) patients: Adriamycin is administered as an IV infusion over a period of 15 minutes at 40 mg/m² on day 2, every 3 weeks (6 cycles); For PET negative (score of 1-3 following Deauville Criteria) patients: Adriamycin is administered as an IV infusion over a period of 15 minutes at 25 mg/m² on day 1 and 15, every 4 weeks (5 cycles)
Drug: Vinblastine — For PET negative (score of 1-3 following Deauville Criteria) patients: Vinblastine is administered as an IV infusion over a period of 15 minutes at 6mg/m² on day 1 and 15, every 4 weeks (5 cycles)
Drug: Dacarbazine — For PET positive (score of 4-5 following Deauville Criteria) patients: Dacarbazine is administered as an IV infusion over a period of 60 minutes at 250 mg/m² on day 3 and 4, every 3 weeks (6 cycles); For PET negative (score of 1-3 following Deauville Criteria) patients: Dacarbazine is administered as an IV infusion over a period of 60 minutes at 375 mg/m² on day 1 and 15, every 4 weeks (5 cycles)
Drug: Etoposide — For PET positive (score of 4-5 following Deauville Criteria) patients: Etoposide is administered as an IV infusion over a period of 60 minutes at 150 mg/m² on day 2,3 and 4, every 3 weeks (6 cycles)
Drug: Cyclophosphamide — For PET positive (score of 4-5 following Deauville Criteria) patients: Cyclophosphamide is administered as an IV infusion over a period of 30 minutes at 1250 mg/m² on day 2, every 3 weeks (6 cycles)
Radiation: Radiation Therapy — Patients with residual lymphoma mass(es) showing metabolic activity of Deauville score 4 or 5 after completion of chemotherapy will be offered consolidation radiotherapy.

SUMMARY:
The main objective of this trial is to assess whether treatment adaptation based on a very early FDG-PET/CT results in improved efficacy while minimizing treatment toxicity in advanced stage Hodgkin Lymphoma (HL) patients treated with brentuximab vedotin (BV)-containing regimens.

DETAILED DESCRIPTION:
This single-arm phase II study investigates the value of early FDG-PET-response adapted BV-based therapy for advanced HL. All patients will receive one cycle of BrAVD followed by an FDG-PET/CT. Patients with a negative early FDG-PET(Deauville score 1-3) will continue with five more BrAVD cycles (total six cycles) while patients with a positive FDG-PET should shift to six cycles of BrECADD.

The hypothesis is that the efficacy will be comparable to the efficacy of BEACOPPesc and BrECADD, while using the intensive chemotherapy regimen only for those patients who do not achieve a negative FDG-PET after one cycle.

The choice to assess the treatment sensitivity by PET after a single cycle of BrAVD is based on results from a recent international multicenter study comparing FDG-PET/CT after one and two cycles of ABVD chemotherapy in HL. There is no reason to suspect that FDG-PET1 should be less prognostic after BrAVD than after ABVD.

With this trial, the investigators believe they can add important information about the optimal treatment of BV-containing first-line treatment for advanced HL, and thus answer important therapeutic questions that are likely to otherwise remain unanswered even after the Echelon-1 and HD21 trials reach mature results. This relatively large single-arm phase II trial of 150 patients will allow a meaningful comparison with the BrAVD and BrECADD regimens based on modified progression-free survival (primary endpoint) and progression-free survival (secondary endpoint) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically proven classical Hodgkin lymphoma;
* Staged by PET with diagnostic-quality CT (i.v. contrast).
* Clinical stages according to Lugano 2014 and based on FDG/PET CT:

  * Stage IIB with large mediastinal mass > 1/3 max transverse diameter thorax and/or extranodal lesion(s)
  * Stage III - IV
* Consent to participation in translational research:
* Archival tumor tissue available (15 blank formalin fixed paraffin embedded tissue samples mounted on APES slides or a tissue block).
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last dose of treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1 percent per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Absence of any medical, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of Progressive Multifocal Leukoencenphalopathy
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
* Sensory or motor peripheral neuropathy greater than or equal to grade 2 according to CTCAE version 4.0
* Any of the following cardiovascular conditions or values:

within 6 months before registration:

* A left-ventricular ejection fraction <50 percent (at registration)
* New York Heart Association (NYHA) Class III or IV heart failure.
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* symptomatic coronary heart disease (stable angina pectoris is allowed)
* severe uncontrolled hypertension within 2 years before registration
* Myocardial infarction
* Patients with poorly controlled diabetes mellitus (HbA1c > 7.5 percent or a fasting blood sugar > 200 mg/dL).
* Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to registration.
* Known HIV infection, chronic active hepatitis C, HBV positivity (HBsAg + patients; HBsAg -/HBcAb+/HBV DNA+ patients).

Note: HBsAg-/HBV DNA - patients are eligible; patients who are seropositive due to vaccination are eligible

* Concomitant or previous malignancies within the past 5 years with the exception of adequately treated carcinoma in situ of the cervix , nonmelanoma skin cancer.
* Previous treatment with anti CD30 antibodies
* Known hypersensitivity to any excipient contained in Brentuximab Vedotin formulation and other study drugs. Refer to Summary Product Characteristics for list of excipients.
* Concurrent anti-cancer treatment or use of any investigational agent(s)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2026-11-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hutchings, Principal Investigator — Past Chair EORTC Lymphoma Group; Wouter Plattel, Principal Investigator — Active Member EORTC Lymphoma Group
Locations (16):
- Belgium (3):
  - ZNA Stuivenberg, Antwerp
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- University Hospitals Copenhagen - Rigshospitalet, Copenhagen, Denmark
- Netherlands (7):
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - Deventer Ziekenhuis, Deventer
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden-Zuid, Leeuwarden
  - Haaglanden Medisch Centrum (HMC) - Haaglanden MC - locatie Antoniushove, Leidschendam
  - Radboudumc - Radboud University Medical Center Nijmegen, Nijmegen
  - Erasmus MC, Rotterdam
- Maria Sklodowska Curie National Institute of Oncology - National Research Institute, Warsaw, Poland
- Instituto Portugues De Oncologia - Francisco Gentil - Centro De Lisboa, Lisbon, Portugal
- National Cancer Institute, Bratislava, Slovakia
- Spain (2):
  - Hospital Duran i Reynals (Institut Catala D'Oncologia), L'Hospitalet de Llobregat
  - Complejo Hospitalario de Navarra, Pamplona

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Patients will receive 1 cycle of BrAVD followed by a PET/CT scan (PET1). Further treatment will be based on the PET1 results scored according to the
  Deauville 5-point score (DS) as follows:
  1. If PET1-negative (DS: 1-3): patients will receive an additional 5 cycles of BrAVD
  2. If PET1-positive (DS: 4-5): patients will switch treatment and receive 6 cycles of BrECADD Radiotherapy will be applied only to patients with residual PET positivity (Deauville 4 or 5) at the end of chemotherapy. Only sites of residual PET positive disease will be irradiated.
Period: Overall Study
Arm/Group | Treatment
Started | 150
Completed | 141
Not Completed | 9
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Poor therapy tolerance, ineligibility, AE, error in treatment administration | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 150
Age, Continuous [Median (Full Range); unit: years] | 32 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 42
  Belgium | 17
  Denmark | 21
  Poland | 2
  Slovakia | 16
  Portugal | 17
  Spain | 35
WHO performance status [Count of Participants; unit: Participants] — 0. Able to carry out all normal activity without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out light work
  2. Ambulatory and capable of all self-care but unable to carry out any work; up and about more than 50% of waking hours
  3. Capable of only limited self-care; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair
  Participants
    0 | 117
    1 | 29
    2 | 4
Histology type [Count of Participants; unit: Participants]
  Nodular sclerosis | 106
  Mixed cellularity | 21
  Lymphocyte depleted | 1
  Lymphocyte rich | 1
  Not otherwise specified | 21
Ann Arbor clinical stage [Count of Participants; unit: Participants] — I: One node or a group of adjacent nodes - Single extranodal lesions without nodal involvement
  II: Two or more nodal groups on the same side of the diaphragm - Stage I or II by nodal extent with limited contiguous extranodal involvement
  III: Nodes on both sides of the diaphragm; nodes above the diaphragm with spleen
  IV: Additional noncontiguous extralymphatic involvement
  The suffix A, B further classifies the stage:
  Category A: The patient does not have B symptoms (fever, weight loss or night sweats).
  Category B: The patient has B symptoms.
  Participants
    IIB | 22
    IIIA | 16
    IIIB | 23
    IVA | 34
    IVB | 55
Any relevant non-malignant medical condition [Count of Participants; unit: Participants]
  No | 44
  Yes | 106
Any history of diabetes mellitus [Count of Participants; unit: Participants]
  No | 148
  Yes | 2
Any history blood hypertension [Count of Participants; unit: Participants]
  No | 136
  Yes | 14
Any malignant medical condition [Count of Participants; unit: Participants]
  No | 149
  Yes | 1

OUTCOME MEASURES:

1. Primary Outcome: Modified Progression-free Survival (mPFS) Rate at 2 Years
Description: Modified PFS (mPFS) is defined as the time interval between the date of treatment start and the date of the first of:
  * Progressive disease (PD)
  * Start of new treatment for Classical Hodgkin Lymphoma (cHL) when not in Complete Response at the end of protocol treatment; in this case, the date of mPFS is the date of the FDG-PET/CT scan at the end of protocol treatment. Switching therapy prior to end of protocol treatment for reasons other than Progressive Disease is not considered an event for mPFS. "End of protocol treatment" refers to completion of the planned protocol treatment with no more than 1 missed cycle, including radiotherapy on PET positive lesions if administered
  * Death due to any cause
Time Frame: 2 years from the date of treatment start
Population: All registered and eligible patients, who started the allocated treatment according to the result of the FDG-PET/CT after 1 cycle of BrAVD, as assessed by central review.
Measure: Number (80% Confidence Interval); unit: Percent probability
Groups:
- Evaluable Population: All registered and eligible patients, who started the allocated treatment according to the result of the FDG-PET/CT after 1 cycle of BrAVD, as assessed by central review.
Arm/Group | Evaluable Population
Number analyzed (Participants) | 145
Percent probability | 89.5 [85.7 to 92.4]

2. Secondary Outcome: Proportion of Patients With a Negative FDG-PET
Description: It will be assessed how many patients have a negative FDG-PET image when taken at the end of their first cycle of BrAVD. The BrAVD cycle lasts 4 weeks.
Time Frame: At day 22 to 23 from start of treatment (day 1 = date of start of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 150
Participants
  Negative | 90
  Positive | 60

3. Secondary Outcome: Progression-free Survival (PFS) Rate at 2 Years
Description: Progression-free survival
Time Frame: 2 years from the date of treatment start
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Evaluable Population
Number analyzed (Participants) | 145
Percent probability | 89.5 [83.3 to 93.6]

4. Secondary Outcome: Overall Survival Rate at 2 Years
Description: Overall survival
Time Frame: 2 years from the date of treatment start
Measure: Number; unit: Percent probability
Arm/Group | Evaluable Population
Number analyzed (Participants) | 145
Percent probability | 100

ADVERSE EVENTS:
Time Frame: Each observed adverse event was to be reported as of 4 weeks within registration until 28 days after start of last cycle of chemotherapy. If radiotherapy given, assessment of adverse events should be done until 8 weeks after completion. Related adverse events should be assessed as of 3 months after the end of treatment until 5 years after end of treatment. All adverse events must be followed until resolution or stabilization. Survival status: assessed until 5 years after end of treatment.
Description: All AEs will be reported in Other section (Serious and non-Serious).
Groups:
- Treatment: Brentuximab Vedotin: For PET positive patients: IV infusion over a period of 30 minutes at 1.8 mg/kg on day 1, every 3 weeks (6 cycles); For PET negative patients: IV infusion over a period of 30 minutes at 1.2 mg/kg on day 1 and 15, every 4 weeks (5 cycles)
  Adriamycin: For PET positive patients: IV infusion over a period of 15 minutes at 40 mg/m² on day 2, every 3 weeks (6 cycles); For PET negative (score of 1-3 following Deauville Criteria) patients: IV infusion over a period of 15 minutes at 25 mg/m² on day 1 and 15, every 4 weeks (5 cycles)
  Vinblastine: For PET negative patients: IV infusion over a period of 15 minutes at 6mg/m² on day 1 and 15, every 4 weeks (5 cycles)
  Dacarbazine: For PET positive patients: IV infusion over a period of 60 minutes at 250 mg/m² on day 3 and 4, every 3 weeks (6 cycles); For PET negative (score of 1-3 following Deauville Criteria) patients: IV infusion over a period of 60 minutes at 375 mg/m² on day 1 and 15, every 4 weeks (5 cycles)
  Etoposide: For PET positive patients: administered as an IV infusion over a period of 60 minutes at 150 mg/m² on day 2,3 and 4, every 3 weeks (6 cycles)
  Cyclophosphamide: For PET positive patients: administered as an IV infusion over a period of 30 minutes at 1250 mg/m² on day 2, every 3 weeks (6 cycles)
  Radiation Therapy: Patients with residual lymphoma mass(es) showing metabolic activity of Deauville score 4 or 5 after completion of chemotherapy will be offered consolidation radiotherapy.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 45/150
Other Adverse Events (participants affected / at risk) | 149/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=150)
ANAEMIA (Blood and lymphatic system disorders) | 4 (7)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 10 (16)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (6)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (2)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
PRINZMETAL ANGINA (Cardiac disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 5 (5)
ILEUS (Gastrointestinal disorders) | 1 (1)
INTESTINAL PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 2 (3)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 3 (3)
MUCOSAL INFLAMMATION (General disorders) | 1 (1)
PYREXIA (General disorders) | 3 (3)
HEPATIC HAEMORRHAGE (Hepatobiliary disorders) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 2 (2)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 3 (3)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 (1)
MENINGITIS (Infections and infestations) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1)
ORAL INFECTION (Infections and infestations) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 5 (5)
PNEUMONIA (Infections and infestations) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
THROMBOPHLEBITIS SEPTIC (Infections and infestations) | 2 (2)
TOOTH ABSCESS (Infections and infestations) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 1 (1)
TUBO-OVARIAN ABSCESS (Infections and infestations) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 2 (3)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
AUTONOMIC NEUROPATHY (Nervous system disorders) | 1 (1)
DEMYELINATING POLYNEUROPATHY (Nervous system disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2)
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 (3)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=150)
ANEMIA (Blood and lymphatic system disorders) | 40 (147)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 14 (23)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 3 (4)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (3)
SINUS TACHYCARDIA (Cardiac disorders) | 7 (7)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1)
MIDDLE EAR INFLAMMATION (Ear and labyrinth disorders) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 4 (4)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 (1)
BLEPHARITIS (Eye disorders) | 1 (1)
DRY EYE (Eye disorders) | 8 (8)
ABDOMINAL PAIN (Gastrointestinal disorders) | 29 (43)
ANAL FISSURE (Gastrointestinal disorders) | 2 (2)
ANAL PAIN (Gastrointestinal disorders) | 1 (1)
BLOATING (Gastrointestinal disorders) | 1 (2)
BURNING FEELING STOMACH (Gastrointestinal disorders) | 1 (1)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 (5)
CONSTIPATION (Gastrointestinal disorders) | 56 (82)
DIARRHEA (Gastrointestinal disorders) | 28 (35)
DRY MOUTH (Gastrointestinal disorders) | 5 (5)
DYSPEPSIA (Gastrointestinal disorders) | 6 (8)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (2)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (3)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 3 (4)
GASTROENTERITIS (Gastrointestinal disorders) | 2 (2)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3)
GASTROINTESTINAL DISORDERS - BLOOD IN STOOL (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL DISORDERS - HEARTBURN (Gastrointestinal disorders) | 1 (4)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1)
GLOSSITIS (Gastrointestinal disorders) | 1 (1)
HEARTBURN (Gastrointestinal disorders) | 1 (1)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 5 (5)
ILEUS (Gastrointestinal disorders) | 1 (1)
MUCOSITIS (OF MOUTH, ESOPHAGUS, STOMACH AND DUODENUM) (Gastrointestinal disorders) | 1 (1)
MUCOSITIS OF MOUTH, ESOPHAGUS, STOMACH AND DUODENDUM (Gastrointestinal disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 24 (39)
NAUSEA (Gastrointestinal disorders) | 64 (126)
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 1 (2)
OBSTIPATION (Gastrointestinal disorders) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 4 (5)
OTHER GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 1 (1)
PYROSIS (Gastrointestinal disorders) | 2 (2)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
REFLUX (Gastrointestinal disorders) | 1 (1)
ROUGH GUM (Gastrointestinal disorders) | 1 (1)
SENSITIVE MOUTH (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (2)
STOMACH PAIN (Gastrointestinal disorders) | 7 (12)
TOOTHACHE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 31 (49)
EDEMA LIMBS (General disorders) | 1 (1)
FATIGUE (General disorders) | 53 (88)
FEVER (General disorders) | 24 (45)
FLU LIKE SYMPTOMS (General disorders) | 5 (6)
GENERAL DISORDERS - WARM-COLD FEELING (General disorders) | 1 (1)
GENERALIZED EDEMA (General disorders) | 2 (2)
INFUSION RELATED REACTION (General disorders) | 1 (1)
IRRITABILITY (General disorders) | 1 (1)
LOCALIZED EDEMA (General disorders) | 3 (3)
MALAISE (General disorders) | 9 (12)
NON-CARDIAC CHEST PAIN (General disorders) | 7 (8)
PAIN (General disorders) | 6 (6)
HEPATIC HEMORRHAGE (Hepatobiliary disorders) | 1 (1)
HEPATIC TOXICITY (Hepatobiliary disorders) | 2 (2)
HEPATITIS VIRAL (Hepatobiliary disorders) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 3 (5)
HYPOGAMMAGLOBULINEMIA (Immune system disorders) | 1 (1)
THYMUS HYPERPLASIA (Immune system disorders) | 1 (1)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1)
BACTEREMIA (Infections and infestations) | 2 (2)
CATHETER RELATED INFECTION (Infections and infestations) | 3 (5)
COVID 19 INFECTION (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 INFECTION (Infections and infestations) | 3 (3)
COVID19 INFECTION (Infections and infestations) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 4 (8)
EYE INFECTION (Infections and infestations) | 1 (1)
FOLLICULITIS (Infections and infestations) | 1 (1)
HERPES SIMPLEX REACTIVATION (Infections and infestations) | 6 (7)
INFECTION (Infections and infestations) | 3 (3)
INFECTION, STAPHYLOCOCCUS HAEMOLYTICUS (Infections and infestations) | 1 (1)
INFECTION, UNKNOWN FOCUS (Infections and infestations) | 2 (6)
INFECTIONS AND INFESTATIONS, OTHER (COVID-19) (Infections and infestations) | 1 (1)
LIP INFECTION (Infections and infestations) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 7 (11)
MENINGITIS (Infections and infestations) | 1 (1)
MOUTH INFECTION (Infections and infestations) | 1 (2)
MUCOSAL INFECTION (Infections and infestations) | 2 (2)
OTITIS MEDIA (Infections and infestations) | 1 (2)
OVARIAN INFECTION (Infections and infestations) | 1 (2)
PAPULOPUSTULAR RASH (Infections and infestations) | 2 (4)
PHARYNGITIS (Infections and infestations) | 6 (7)
PHLEBITIS INFECTIVE (Infections and infestations) | 1 (1)
PNEUMOCYSTIS JIROVECI PNEUMONIA INFECTION (Infections and infestations) | 1 (3)
RHINITIS INFECTIVE (Infections and infestations) | 2 (2)
SEPSIS (Infections and infestations) | 2 (4)
SEPTIC THROMBOPHLEBITIS (Infections and infestations) | 1 (3)
SHINGLES (Infections and infestations) | 3 (3)
SINUSITIS (Infections and infestations) | 2 (2)
SKIN INFECTION (Infections and infestations) | 3 (3)
SMALL INTESTINE INFECTION (Infections and infestations) | 1 (1)
SUSPECTED PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 (2)
SUSPICIOUS INFECTION (Infections and infestations) | 1 (1)
THRUSH (Infections and infestations) | 6 (7)
TONSILLITIS (Infections and infestations) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 7 (9)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 7 (8)
UPPER RESPIRATORY TRACT INFECTION DUE TO INFLUENZA A (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5)
VAGINAL INFECTION (Infections and infestations) | 5 (5)
WOUND INFECTION (Infections and infestations) | 1 (1)
ZOSTER (Infections and infestations) | 1 (2)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 5 (7)
PAIN PICC KATHETER (Injury, poisoning and procedural complications) | 1 (1)
PAINFUL VEIN AFTER INFUSION (Injury, poisoning and procedural complications) | 1 (1)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 16 (22)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 9 (9)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 5 (5)
CARBON MONOXIDE DIFFUSING CAPACITY DECREASED (Investigations) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 2 (2)
FORCED EXPIRATORY VOLUME DECREASED (Investigations) | 1 (1)
GGT INCREASED (Investigations) | 2 (3)
LYMPHOCYTE COUNT DECREASED (Investigations) | 6 (7)
NEUTROPHIL COUNT DECREASED (Investigations) | 55 (149)
PLATELET COUNT DECREASED (Investigations) | 17 (85)
TRANSAMINITIS (Investigations) | 1 (3)
WEIGHT GAIN (Investigations) | 12 (23)
WEIGHT LOSS (Investigations) | 17 (32)
WHITE BLOOD CELL DECREASED (Investigations) | 18 (60)
WHITE BLOOD CELL INCREASED (Investigations) | 1 (1)
WHITE BLOOD CELLS INCREASED (Investigations) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 16 (26)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 8 (12)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1)
TUMOR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 (9)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 (22)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 27 (42)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
FATIGUE IN ARMS (Musculoskeletal and connective tissue disorders) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (4)
INFLAMMATION OF TENDONS (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 4 (4)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 23 (34)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5)
OTHER, HEAVY ARMS AND LEGS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN BACK/HIPS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 (9)
PAIN RIBS/HIP (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN, GROIN (Musculoskeletal and connective tissue disorders) | 1 (1)
STERNUM DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 (1)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ANOSMIA (Nervous system disorders) | 1 (1)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 3 (3)
DIZZINESS (Nervous system disorders) | 11 (13)
DYSGEUSIA (Nervous system disorders) | 20 (28)
DYSPHASIA (Nervous system disorders) | 1 (1)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 16 (25)
MEMORY IMPAIRMENT (Nervous system disorders) | 2 (2)
PARESTHESIA (Nervous system disorders) | 16 (18)
PERIPHERAL AUTONOMIC NEUROPATHY (Nervous system disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 30 (42)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 79 (149)
SENSITIVE MOTOR SYNDROME (Nervous system disorders) | 1 (1)
SENSORY AND MOTOR POLYNEUROPATHY (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2)
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 1 (1)
VEGETATIVE NEUROPATHY (Nervous system disorders) | 1 (1)
AGITATION (Psychiatric disorders) | 2 (3)
ANXIETY (Psychiatric disorders) | 6 (6)
INSOMNIA (Psychiatric disorders) | 26 (31)
IRRITABILITY (Psychiatric disorders) | 1 (1)
PSYCHIATRIC DISORDERS - EMOTIONAL DISTRESS (Psychiatric disorders) | 3 (3)
RESTLESSNESS (Psychiatric disorders) | 2 (2)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 3 (3)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 2 (3)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1)
URINE DISCOLORATION (Renal and urinary disorders) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 3 (4)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PREMATURE MENOPAUSE (Reproductive system and breast disorders) | 3 (4)
SCROTAL PAIN (Reproductive system and breast disorders) | 1 (2)
TESTICULAR PAIN (Reproductive system and breast disorders) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (16)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 16 (20)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
EXTRINSIC ALLERGIC ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 5 (7)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMPYEMA (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PULMONARY TOXICITY WITH REDUCT OF CARB MONOX DIFFUSING CAPAC (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 5 (5)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 5 (5)
ACNE (Skin and subcutaneous tissue disorders) | 1 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 16 (22)
BODY ODOR (Skin and subcutaneous tissue disorders) | 1 (1)
CUTANEOUS ABSCESS (Skin and subcutaneous tissue disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 8 (8)
ECZEMA (Skin and subcutaneous tissue disorders) | 4 (4)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1)
EXANTHEM (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 11 (11)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 11 (12)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 11 (14)
RIGHT AXILLARY HIDRADENITIS SUPPURATIVA (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - EASILY GETS WOUNDS (Skin and subcutaneous tissue disorders) | 1 (2)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - SENSITIVE SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS- SKIN IRRITATION ANUS (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
SWEET SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
FLUSHING (Vascular disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 4 (4)
HYPERTENSION (Vascular disorders) | 20 (53)
HYPOTENSION (Vascular disorders) | 1 (1)
PHLEBITIS (Vascular disorders) | 2 (2)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 1 (1)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT03517137/Prot_SAP_000.pdf